CLINICAL TRIAL: NCT01003834
Title: Computer vs Therapist-Delivered Brief Interventions for Substance Use in Primary Care
Brief Title: Computerized Screening, Brief Intervention, and Referral to Treatment in Primary Care
Acronym: SBIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SBIRTVCU; R01DA026091 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Substance Use Disorder
Keywords: substance use; drug use; drug abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Placebo Comparator): Screening only
  Interventions: Behavioral: Computerized health screening
- Assessment (Active Comparator): Screening plus assessment
  Interventions: Behavioral: Computerized health screening; Behavioral: Computerized assessment
- Computer Intervention (Experimental): Screening, assessment, and computer-delivered intervention
  Interventions: Behavioral: Computerized brief intervention; Behavioral: Computerized health screening; Behavioral: Computerized assessment
- Therapist Intervention (Active Comparator): Screening, Assessment, and therapist-delivered intervention
  Interventions: Behavioral: Computerized health screening; Behavioral: Computerized assessment; Behavioral: Therapist-delivered motivational intervention

INTERVENTIONS:
Behavioral: Computerized brief intervention — Intervention based on Motivational Interviewing technique
  Arms: Computer Intervention
Behavioral: Computerized health screening — Behavioral intervention
Behavioral: Computerized assessment — Behavioral intervention
  Arms: Assessment; Computer Intervention; Therapist Intervention
Behavioral: Therapist-delivered motivational intervention — Behavioral intervention
  Arms: Therapist Intervention

SUMMARY:
This is a randomized, controlled clinical trial to evaluate the effect of a computerized screening, assessment, and brief intervention on substance use in patients recruited from a primary care clinic. Study participants will be assigned to one of the following 4 study groups: computerized health screening alone (standard care) (SC); computerized assessment-only intervention (CA); computerized assessment followed by a computer-directed motivational intervention (CACI); or computerized assessment followed by a therapist-delivered motivational intervention (CATI). Data regarding substance use, medical and psychosocial functioning, and economic outcomes will be collected.

The investigators hypothesize that patients randomized to CACI and CATI will be more likely to report drug abstinence at the 3-month follow-up visit and will show greater reductions in drug use at 1, 3 and 6 months follow-up than patients assigned to CA or SC. Similarly, patients in the CACI and CATI groups will report greater reductions in HIV risk behaviors, lower rates of medical and psychosocial problems, and increased economic gains at the 6-month follow-up. In addition, patients in the assessment only intervention (CA) will have outcomes superior to those found for SC patients. A cost-effectiveness analysis will also be done comparing economic costs associated with CA, CACI and CATI and their relationship to substance use reductions and related improvements in medical and psychosocial outcomes at the 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* Primary care clinic patient

Exclusion Criteria:

* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Substance use | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States